CLINICAL TRIAL: NCT02266303
Title: The Effect of a Checklist on the Education of Simulated Patients During Insulin Initiation: a Randomized Controlled Trial
Brief Title: The Effect of a Checklist on the Education of Simulated Patients During Insulin Initiation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UWestIndies
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Insulin Checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With checklist (Experimental): Doctors will initiate insulin with the aid of a checklist
  Interventions: Other: Insulin Start-up Checklist
- Without checklist (No Intervention): Doctors will initiate insulin without the use of the checklist

INTERVENTIONS:
Other: Insulin Start-up Checklist — The checklist is a simple A4 size, two sided, document. Eleven checklist items covering twenty-one key educational points are of the front. Images illustrating the process of using a syringe to draw up insulin from a vial as well as injection sites (for children, adults and pregnant women) are on the back.
  Arms: With checklist

SUMMARY:
The increasing prevalence of diabetes is associated with increased insulin use. In developing countries it is frequently necessary to use insulin, with the needle and syringe method of administration being the cheapest approach. Competence of health care professionals is required to safely initiate insulin. The investigators will evaluate whether using a checklist during insulin initiation with a needle and syringe, can improve the safety and efficacy of its use.

DETAILED DESCRIPTION:
Introduction The prevalence of type 2 diabetes mellitus is increasing worldwide with a disproportionate increase in developing countries [1]. The burden is tremendous in developing countries, where the greatest increases are expected over time. For example, the prevalence of diabetes in adults in the North American and the Caribbean region is expected to increase by 37% in 2035. However, the increase in Africa and South and Central America over the same time period is expected to be 109% and 60% respectively[1].

This crisis is further compounded by the demand on financial resources placed by the high cost of care. Estimated costs of diabetes care reached $239.2 billion United Sates Dollars (USD) in 2013 in The North American and Caribbean region[2]. Abdulkadri et al estimated the economic cost of both diabetes and hypertension in four Caribbean countries (Barbados, Jamaica, Trinidad and Tobago and The Bahamas) in 2001 to be 753 million USD per year[3].

The management of type 2 diabetes has evolved from an algorithmic approach[4], towards individualized care[5, 6], but affordability limits treatment options in many developing countries. The evolution was driven by the increased availability of drugs used in diabetes treatment. However, drug availability has not equally penetrated the developed and developing world due to cost. Insulin in its cheapest forms (animal or human administered by a syringe) therefore remains critical in the management of diabetes in the developing world given its lower cost and greater efficacy. For example, Dipeptidyl peptidase-4 inhibitors cost approximately twice that of a month's supply of syringe delivered, intermediate human insulin, at a dose of 40 units daily. However, the potential reduction of HbA1C is 0.5-0.8% with DPP-4 inhibitors but as much as 3.5% with insulin titration[7]. Even in the developed world, the global financial crisis may result in similar shifts in lower income groups.

It is therefore critical for healthcare professionals to know how to safely initiate insulin. For insulin to be safely used, particularly by the needle and syringe method, healthcare professionals must adequately educate patients in a number of areas. These areas include side effects, drawing up and administration of insulin, and the recognition and treatment of hypoglycaemia. Given the complexity of the task all areas may not be recalled by health care professionals during a patient encounter.

The task of insulin initiation can be simplified through the use of a checklist. Ely and colleagues believe that checklists are an alternative to reliance on memory and reduce diagnostic errors[8]. Depending solely on recall is likely to open the gateway for omissions, particularly given that there is poor representation of structured teaching on insulin initiation during undergraduate medical training. An insulin initiation checklist can also simultaneously provide education for the healthcare professionals using insulin.

Using human patient simulation we will evaluate the potential safety benefit of using a checklist for insulin initiation by the syringe method. Human patient simulation allows the assessment of clinical knowledge and skills without exposing individuals to risk.

Research hypothesis (alternate) The use of a checklist during insulin initiation via needle and syringe, can improve patient education on safe and effective insulin use.

Methods Trial design

We will conduct a randomized controlled study. Participants will complete the simulation on insulin initiation twice. Participants will be randomly assigned to the following groups and each simulation will be separated by a 5 to 10-minute period as outlined below:

Group 1 (intervention group) - Participants will complete the simulation without the checklist. They will then be introduced to the checklist and allowed up to ten minutes to review it. They will subsequently repeat the simulation while using the checklist.

Group 2 (control group) - Participants will complete the simulation initially without the checklist, as in group 1. They will then be allowed up to ten minutes to reflect on the exercise. They will subsequently repeat the simulation exercise, but again without the availability of the checklist.

The study design will attempt to ensure any improvements identified in association with the checklist can be attributed to its use and not to a learning effect or previous skills.

Performance during each simulation will be assessed with the aid of a check sheet. Educational tasks will be listed on this sheet under the headings of 'Side Effects', 'Hypoglycemia', 'Drawing up insulin', 'Administration of insulin' and 'Other'. Tick boxes will be used to check off whether tasks are performed adequately, inadequately or not at all. Each task will have brief notes on what constitute adequate performance.

The Checklist The checklist was developed by a taskforce. The group consisted of 11 individuals; a layperson, a pharmacist, two dietitians, two diabetes educators, a podiatrist, a diabetes specialist nurse, a pediatrician and two diabetologists. The process was lead by the pharmacist, diabetes specialist nurse and one of the diabetologists. The first version was created by the three healthcare professionals leading the process, however the final version was achieved through four iterative cycles of feedback and re-design.

The aim was to develop a simple A4 size, two sided, document that could be easily copied. Eleven checklist items were agreed upon which covered twenty-one key educational points for safe and effective insulin initiation. These educational points fell under four themes - insulin side effects, recognition and treatment of hypoglycemia, drawing up insulin with a syringe, and administration of insulin.

Images illustrating the process of using a syringe to draw up insulin from a vial as well as injection sites (for children, adults and pregnant women) were included at the back. There was also space provided for documentation of the client's name and registration number, insulin type and when it should be taken, medications to be stopped, and the date and signature of the facilitator.

Setting and simulation The interns will be asked to complete the simulation in the Clinical Skills Building of The University of the West Indies. Established practitioners will have the simulation carried out at their offices. During the simulation an actor/actress will require education on the use and administration of insulin via a needle and syringe. The participant will be given the equipment (insulin syringes and needles, injection pad and insulin) and instructions for the exercise, which will include the clinical scenario.

Analysis Chi-squared analyses will establish whether the intervention and control groups are equivalent with respect to demographic variables (age, gender, etc). The paired t-test will determine differences between pair measurements of performance within groups, and the student t-test between groups. If the necessary assumptions do not apply, the Wilcoxon ranked sum test and Wilcoxon signed- rank test will be used respectively. Associations between demographic variables and outcome variables will be determined using Pearson's correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Registered General Practitioners in 2014, by the Barbados Medical Council, including those just recently completing supervised internship in June 2014.

Exclusion Criteria:

* Practitioners not registered with the Barbados Medical Council in 2014

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The total number of educational points addressed for the safe and effective use of insulin (of the possible 21 identified). | 5 months

SECONDARY OUTCOMES:
The number of educational points addressed under each of the four themes of insulin side effects, hypoglycemia, drawing up and administering insulin. | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Cave Hill Campus, Bridgetown, Saint Michael, Barbados

REFERENCES:
- [Background] 1. Guariguata, L. and F. International Diabetes, IDF diabetes atlas. 6th ed. 2013, Brussels: International Diabetes Federation. 159 p.
- [Background] Yisahak SF, Beagley J, Hambleton IR, Narayan KM; IDF Diabetes Atlas. Diabetes in North America and the Caribbean: an update. Diabetes Res Clin Pract. 2014 Feb;103(2):223-30. doi: 10.1016/j.diabres.2013.11.009. Epub 2013 Dec 1. PMID 24321468
- [Background] 3. Abdulkadri, A.O., et al., ECONOMIC BURDEN OF DIABETES AND HYPERTENSION IN CARICOM STATES. Social and Economic Studies, 2009. 58(3/4): p. 175.
- [Background] Bailey T. Options for combination therapy in type 2 diabetes: comparison of the ADA/EASD position statement and AACE/ACE algorithm. Am J Med. 2013 Sep;126(9 Suppl 1):S10-20. doi: 10.1016/j.amjmed.2013.06.009. PMID 23953074
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] Qaseem A, Humphrey LL, Sweet DE, Starkey M, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Oral pharmacologic treatment of type 2 diabetes mellitus: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2012 Feb 7;156(3):218-31. doi: 10.7326/0003-4819-156-3-201202070-00011. PMID 22312141
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Ely JW, Graber ML, Croskerry P. Checklists to reduce diagnostic errors. Acad Med. 2011 Mar;86(3):307-13. doi: 10.1097/ACM.0b013e31820824cd. PMID 21248608
- [Derived] Taylor CG Jr, Bynoe K, Worme A, Hambleton I, Atherley A, Husbands A, Unwin N. A checklist that enhances the provision of education during insulin initiation simulation: a randomized controlled trial. Diabet Med. 2016 Sep;33(9):1204-10. doi: 10.1111/dme.12956. Epub 2015 Oct 16. PMID 26337285